CLINICAL TRIAL: NCT02153021
Title: New Therapeutic Perspectives in Obesity
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Nivaldo Antonio Parizotto, PhD, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 231.286
Record Dates: First submitted 2014-04-28; First posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Obesity;
Keywords: anthropometric parameters;; biochemical parameters;; inflammatory markers; neuropeptide markers; phototherapy
MeSH Terms: conditions — Obesity | interventions — Phototherapy; Lasers; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Placebo Comparator): alimentation information: a nutritionist provides nutritional orientation; exercise training: 3 days by week the patients will have specific sessions of resistance training (30 minutes) and aerobic training (30 minutes); phototherapy: all patients will received application of phototherapy after exercise session. The phototherapy will be applicated in abdominal and dorsal circumference/ quadriceps and biceps femoral. In Sham group,the equipment will be off.
- Phototherapy (Active Comparator): phototherapy: all patientes will received application of phototherapy after exercise session. The phototherapy will be applicated in abdominal and dorsal circumference/ quadriceps and biceps femoral.
  Type Ga-Al-As Wavelength 808nm Frenquency Continue wave Optical output 100mW Spot diameter 0.6mm Power density 60W/cm2 Energy per minute 6J/point Number of Points 64points Total energy delivered 48J
  Interventions: Radiation: Phototherapy

INTERVENTIONS:
Radiation: Phototherapy — phototherapy: all patientes will received application of phototherapy after exercise session. The phototherapy will be applicated in abdominal and dorsal circumference/ quadriceps and biceps femoral.
  Type Ga-Al-As Wavelength 808nm Frenquency Continue wave Optical output 100mW Spot diameter 0.6mm Power density 60W/cm2 Energy per minute 6J/point Number of Points 64points Total energy delivered 48J
  Other Names: laser; lasertherapy; low-level laser therapy
  Arms: Phototherapy

SUMMARY:
Obesity is a chronic disease of increasing prevalence, being currently considered a global epidemic, including children, adolescents, adults and the elderly of different nationalities and ethnicities, socioeconomic levels, education levels. Non-pharmacological therapeutic interventions, such as physical exercise and fitness healthy eating strategies seem to be increasingly studied and recommended for healthy weight loss. In addition, therapies that can complement the effect of exercise and diet for reducing body weight are considerate important strategies. Thus, experimental evidence shows that the use of laser therapy combined with exercise swimming was effective in controlling the lipid profile, reducing the mass of adipose tissue, suggesting increased metabolic activity and changes in lipid metabolism.

To investigate the effect of the use of therapeutic laser when associated to exercise like response to new therapy for weight loss and decrease of dyslipidemias levels.

DETAILED DESCRIPTION:
Methods:

During 20 weeks, each patients will receive 3 session of exercise with duration of 1 hour. Each session of exercise will composed of aerobic exercise and resistence exercise. After training session, each patient will receive application of phototherapy during 16 minutes. The protocol of phototherapy appplication is described in link "interventions"

ELIGIBILITY:
Inclusion Criteria:

* volunteers aged 20-40 years with a body mass index (BMI) ≥ 30 above, of both genders with primary obesity;

Exclusion Criteria:

* The criteria for inclusion are volunteers who use contraceptive use, cortisone, anti-epileptic drugs, history of kidney and heart disease, alcohol abuse, smoking, use of supplemental vitamins or secondary diagnosis of obesity.

After the pre-selection in the initial interview, the volunteers who contemplate all the inclusion criteria will be referred for clinical evaluation with an interdisciplinary health team and the electrocardiogram stress test to verify the release of the practice of physical exercises proposed by the project .

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Anthropometric measure | the measure occur up to 20 weeks
  Weight body: this measure would occurs during each week.
anthropometric parameter | the measure occur up to 20 weeks
  total body fat: this measure would occurs during each week
anthropometric parameter | the measure occur up to 20 weeks
  visceral body fat: this measure would occurs during each week
anthropometric parameter | the measure occur up to 20 weeks
  total muscle

SECONDARY OUTCOMES:
Primary biochemical analyzes | the measures occur up to 20 weeks
  The primary biochemical: glicemic variables (glucose and insulin)
Primary biochemical analyzes | the measure occur up to 20 weeks
  the lipids variables (total cholesterol; triglycerides; low density lipoprotein; very low density lipoprotein; high density lipoprotein)

OTHER OUTCOMES:
measure of neuropeptide | measures up to 20 weeks
  neuropeptides variables: neuropeptide Y (NPY); agouti-related peptide (agRP); melanotropic hormone (MCH); Leptine; alpha melanocyte stimulating (alpha MSH); Pro-opiomelanocortin (POMC); Cocaine-Amphetamine-Regulated Transcript (CART);
measure of interleukines and citokines | the measure occur up to 20 weeks
  interleukines and citokines variables: iL-1; iL-4; iL-6; iL-10; c reactive protein.

CONTACTS AND LOCATIONS:
Overall Officials: Nivaldo A Parizotto, PhD, Principal Investigator — Universidade Federal de Sao Carlos
Locations (1):
- Unversidade Federal de São Carlos, São Carlos, São Paulo, Brazil